CLINICAL TRIAL: NCT04521621
Title: A Phase 1b/2 Clinical Study of Intratumoral Administration of V937 in Combination With Pembrolizumab (MK-3475) in Participants With Advanced/Metastatic Solid Tumors
Brief Title: A Study of Gebasaxturev (V937) in Combination With Pembrolizumab (MK-3475) in Participants With Advanced/Metastatic Solid Tumors (V937-013)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Business Reasons
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: V937-013; V937-013 (Other: MSD); jRCT2033200191 (Registry Identifier: jRCT); 2020-001908-42 (EudraCT Number)
Record Dates: First submitted 2020-08-17; First posted 2020-08-20 (Actual); Results first posted 2024-08-07 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Neoplasm Metastasis
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Death-Ligand 1 (PDL1, PD-L1)
MeSH Terms: conditions — Neoplasm Metastasis; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Part 1, Cohort A: Triple-Negative Breast Cancer (Experimental): This arm will enroll participants with triple-negative breast cancer (TNBC) solid tumors. Participants receive 3 X 10^8 50% tissue culture infectious dose (TCID50) of gebasaxturev intratumorally for 8 cycles, and pembrolizumab intravenously for a maximum of 35 cycles. Cycle 1 is 28 days, and cycles 2-35 are 21 days.
  Interventions: Biological: Gebasaxturev; Drug: Pembrolizumab
- Part 1, Cohort B: Head and Neck Squamous Cell Carcinoma (Experimental): This arm will enroll participants with head and neck squamous cell carcinoma (HNSCC) solid tumors. Participants receive 3 X 10^8 TCID50 of gebasaxturev intratumorally for 8 cycles, and pembrolizumab intravenously for a maximum of 35 cycles. Cycle 1 is 28 days, and cycles 2-35 are 21 days.
  Interventions: Biological: Gebasaxturev; Drug: Pembrolizumab
- Part 1, Cohort C: Cutaneous Squamous Cell Carcinoma (Experimental): This arm will enroll participants with cutaneous squamous cell carcinoma (cSCC) solid tumors. Participants receive 3 X 10^8 TCID50 of gebasaxturev intratumorally for 8 cycles, and pembrolizumab intravenously for a maximum of 35 cycles. Cycle 1 is 28 days, and cycles 2-35 are 21 days.
  Interventions: Biological: Gebasaxturev; Drug: Pembrolizumab
- Part 2 Dose Level 1, Solid Tumors + Liver Metastases (Experimental): This arm will enroll participants with solid tumors with liver metastases. Participants receive 3 X 10^7 TCID50 of gebasaxturev intratumorally for 8 cycles, and pembrolizumab intravenously for a maximum of 35 cycles. Cycle 1 is 28 days, and cycles 2-35 are 21 days.
  Interventions: Biological: Gebasaxturev; Drug: Pembrolizumab
- Part 2 Dose Level 2, Solid Tumors + Liver Metastases (Experimental): This arm will enroll participants with solid tumors with liver metastases. Participants receive 1 X 10^8 TCID50 of gebasaxturev intratumorally for 8 cycles, and pembrolizumab intravenously for a maximum of 35 cycles. Cycle 1 is 28 days, and cycles 2-35 are 21 days.
  Interventions: Biological: Gebasaxturev; Drug: Pembrolizumab
- Part 2 Dose Level 3, Solid Tumors + Liver Metastases (Experimental): This arm will enroll participants with solid tumors with liver metastases. Participants receive 3 X 10^8 TCID50 of gebasaxturev intratumorally for 8 cycles, and pembrolizumab intravenously for a maximum of 35 cycles. Cycle 1 is 28 days, and cycles 2-35 are 21 days.
  Interventions: Biological: Gebasaxturev; Drug: Pembrolizumab
- Part 2, Cohort D: Hepatocellular Carcinoma (HCC) (Experimental): This arm will enroll participants with hepatocellular carcinoma (HCC) solid tumors. Participants receive the gebasaxturev recommended phase 2 dose (RP2D) intratumorally for 8 cycles, and pembrolizumab intravenously for a maximum of 35 cycles. Cycle 1 is 28 days, and cycles 2-35 are 21 days.
  Interventions: Biological: Gebasaxturev; Drug: Pembrolizumab
- Part 2, Cohort E: Gastric Carcinoma (Experimental): This arm will enroll participants with gastric carcinoma solid tumors. Participants receive the gebasaxturev recommended phase 2 dose (RP2D) intratumorally for 8 cycles, and pembrolizumab intravenously for a maximum of 35 cycles. Cycle 1 is 28 days, and cycles 2-35 are 21 days.
  Interventions: Biological: Gebasaxturev; Drug: Pembrolizumab

INTERVENTIONS:
Biological: Gebasaxturev — Participants receive gebasaxturev intratumorally for 1 28-day cycle followed by 7 21-day cycles.
  Other Names: Coxsackievirus A21 (CVA21); Formerly known as CAVATAK®; CAV21; V937
Drug: Pembrolizumab — Participants receive pembrolizumab intravenously for 1 28-day cycle followed by 34 21-day cycles.
  Other Names: MK-3475; KEYTRUDA®

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and efficacy in participants with advanced/metastatic or recurrent malignancies who receive gebasaxturev (V937) in combination with pembrolizumab (MK-3475). The primary objective for Part 1 is to evaluate the objective response rate, and the primary objective for Part 2 is to determine the safety and tolerability of gebasaxturev administered in combination with pembrolizumab. With Amendment 4, this study will be terminated once all participants who have completed or discontinued gebasaxturev treatment and are only receiving pembrolizumab may be enrolled in a pembrolizumab extension study, if available, to continue pembrolizumab monotherapy for up to 35 cycles from first pembrolizumab dose on V937-013.

ELIGIBILITY:
Inclusion Criteria:

* Locally-advanced disease that is not amenable to surgery or radiation, or Stage IV advanced/metastatic solid tumor malignancies
* Histologically- or cytologically-confirmed diagnosis of an advanced/metastatic solid tumor.
* Measurable disease by RECIST 1.1 criteria as assessed by investigator. Target lesions in a previously irradiated area will be considered measurable if progression has been demonstrated in such lesions
* Submitted a baseline tumor sample for analysis. Participants enrolling in Part 2 Cohorts D-F may enroll without submitting a tumor sample if all other enrollment criteria are met.
* Performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale obtained within 72 hours prior to the first dose of study intervention
* If participant has known human immunodeficiency virus (HIV)-positive disease, participant must have well-controlled HIV on antiretroviral therapy (ART), per study criteria.
* Adequate organ function
* Male participants are eligible to participate if they agree to the following during the intervention period and for at least 120 days: Be abstinent from heterosexual intercourse as their preferred and usual lifestyle and agree to remain abstinent, OR must agree to use contraception unless confirmed to be azoospermic.
* Female participants are eligible to participate if not pregnant or breastfeeding, and at least one of the following conditions applies:

  * Is not a woman of childbearing potential (WOCBP)
  * Is a WOCBP and using a contraceptive method that is highly effective, or be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis), during the intervention period and for at least 120 days after the last dose of study intervention.
* Contraceptive use by women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* Part 1, All Cohorts: participants must have at least one injectable lesion amenable to injection and/or biopsy.
* Part 1, Cohort A:

  * Locally recurrent, inoperable OR metastatic breast cancer treated with at least 1 prior line of therapy in the metastatic setting with skin involvement and/or subcutaneous lesions or accessible lymph nodes amenable to local injection. An exception would be allowed for participants who are not eligible to receive chemotherapy.
  * Diagnosis of triple-negative breast cancer (estrogen receptor, progesterone receptor, and HER2-receptor negative status)
* Part 1, Cohort B:

  * Histologically confirmed advanced or metastatic head and neck squamous cell carcinoma (HNSCC) of the oral cavity, oropharynx, hypopharynx, and/or larynx considered incurable and/or treated with no more than 1 previous line of therapy
  * Tumors must be PD-L1+
  * Documentation of HPV status for oropharyngeal cancers. Other HNSCC subtypes may submit HPV testing, but is not required.
* Part 1, Cohort C:

  * Histologically confirmed cutaneous squamous cell carcinoma (cSCC) as the primary site of malignancy
  * Recurrent/metastatic disease only: Has metastatic disease defined as disseminated disease distant from the initial/primary site of diagnosis and/or with a history of locally-recurrent disease previously treated with surgery and/or radiotherapy, which is now incurable
  * Locally-advanced disease only: Must be ineligible for surgical resection per study criteria, and must have received prior radiation therapy to the index site or deemed ineligible for radiation therapy
* Part 2, Solid Tumors+Liver Metastases Dose Level 1-3 arms:

  * Histologically-confirmed advanced/metastatic solid tumor that has progressed on all treatment known to confer clinical benefit
  * Metastatic liver lesion(s) not exceeding one-third of the total liver volume AND a minimum of one injectable liver lesion
* Part 2, Cohort D:

  * Advanced hepatocellular carcinoma (HCC) following progression on, or intolerance to, sorafenib or lenvatinib with no curative options
  * Diagnosis of HCC confirmed by radiology, histology, or cytology
  * Child-Pugh Class A score
  * If a participant has a history of hepatitis C virus (HCV) infection, then the participant must have been successfully treated for this condition
  * Controlled (treated) hepatitis B participants will be allowed if they meet protocol-specified criteria
  * Participants who are anti-hepatitis B core (HBc) positive, negative for hepatitis B surface antigen (HBsAg), negative or positive for anti-hepatitis B surface (HBs), and who have an HBV viral load under 100 IU/mL, do not require HBV anti-viral prophylaxis
* Part 2, Cohort E:

  * Histologically- or cytologically-confirmed diagnosis of locally advanced, unresectable or metastatic gastric or gastroesophageal junction (GEJ) adenocarcinoma
  * Received at least one prior line of therapy that includes a platinum/fluoropyrimidine doublet or triplet regimen
  * Had proven clinical progression 6 months following (or during) last dose of adjuvant or neo-adjuvant therapy
  * Human epidermal growth factor receptor 2 (HER2) negative status; or, those with HER2 positive status AND documented disease progression on a prior regimen containing trastuzumab

Exclusion Criteria:

* Chemotherapy, definitive radiation, or biological cancer therapy within 4 weeks (2 weeks for palliative radiation) prior to first dose of study intervention, or has not recovered to Common Terminology Criteria for Adverse Events (CTCAE) Grade 1 or better
* If major or minor surgery was performed at/near the area being considered for injection, participant must be recovered from toxicity and/or complications of intervention
* If participant has had injection or radiation therapy, participant must be recovered from toxicity and/or complications of intervention
* History of second malignancy, unless potentially curative treatment has been completed with no further evidence of disease for ≥5 years.
* Known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Participants with treated brain metastases may participate if lesions are radiologically stable.
* Active infection requiring therapy, except HIV criteria as stated above, and HBV and HCV criteria for HCC cohort as stated above
* History of interstitial lung disease
* History of noninfectious pneumonitis requiring active steroid therapy or ongoing pneumonitis
* Active autoimmune disease that required systemic treatment in the past 2 years except vitiligo or resolved childhood asthma/atopy
* Known Hepatitis B or C infections or known to be positive for HBsAg/HBV deoxyribonucleic acid (DNA) or Hepatitis C Antibody or ribonucleic acid (RNA)
* History of Kaposi's sarcoma and/or Multicentric Castleman's Disease
* Known hypersensitivity to gebasaxturev and/or pembrolizumab or any of their excipients
* Received prior therapy with anti-programmed cell death protein-1 (anti-PD-1), anti-programmed cell death-ligand 1 (anti-PD-L1) agents, Talimogene Laherparepvec (T-VEC), or any other oncolytic virus therapies
* Received a live or live-attenuated vaccine within 30 days prior to first dose of study intervention. Administration of killed vaccines is allowed.
* Pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of study intervention
* Part 2, Cohort D:

  * Has had esophageal or gastric variceal bleeding within the last 6 months
  * Has had clinically diagnosed hepatic encephalopathy in the 6 months prior to initiation of study intervention
* Part 2, Cohort E:

  * Squamous cell or undifferentiated gastric cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2020-10-28 (Actual); Primary Completion 2023-07-25 (Actual); Study Completion 2023-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (29):
- United States (2):
  - John Theurer Cancer Center ( Site 0004), Hackensack, New Jersey
  - Providence Portland Medical Center ( Site 0001), Portland, Oregon
- Canada (2):
  - Princess Margaret Cancer Centre ( Site 0031), Toronto, Ontario
  - Centre Hospitalier de l Universite de Montreal - CHUM ( Site 0032), Montreal, Quebec
- France (3):
  - Centre Hospitalier Lyon-Sud ( Site 0055), Pierre-Bénite, Auvergne-Rhône-Alpes
  - Hopital La Timone ( Site 0051), Marseille, Bouches-du-Rhone
  - Gustave Roussy ( Site 0053), Villejuif, Val-de-Marne
- Germany (2):
  - Universitaetsklinikum Heidelberg-Nationales Centrum für Tumorerkrankungen ( Site 0172), Heidelberg, Baden-Wurttemberg
  - Universitaetsklinikum Tuebingen ( Site 0171), Tübingen, Baden-Wurttemberg
- Orszagos Onkologiai Intezet ( Site 0070), Budapest, Hungary
- Israel (3):
  - HaEmek Medical Center ( Site 0071), Afula
  - Hadassah Medical Center. Ein Kerem ( Site 0072), Jerusalem
  - Sourasky Medical Center ( Site 0073), Tel Aviv
- Istituto Europeo di Oncologia IRCCS-Divisione di Sviluppo di Nuovi Farmaci per Terapie Innovative (, Milan, Italy
- National Cancer Center Hospital East ( Site 0166), Kashiwa, Chiba, Japan
- Norway (2):
  - Helse Bergen HF - Haukeland Universitetssykehus ( Site 0162), Bergen, Hordaland
  - Oslo Universitetssykehus Radiumhospitalet ( Site 0161), Oslo
- Clinica San Gabriel ( Site 0097), Lima, Peru
- Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - P-Oddzial Badan Wczesnych Faz ( Site 0181, Warsaw, Masovian Voivodeship, Poland
- Portugal (2):
  - Centro Hospitalar Universitário Lisboa Norte, E.P.E. - Hospital de Santa Maria ( Site 0192), Lisbon, Lisbon District
  - Instituto Português de Oncologia do Porto Francisco Gentil, EPE ( Site 0191), Porto
- Spain (2):
  - Hospital Universitari Vall d Hebron ( Site 0121), Barcelona
  - Clinica Universitaria de Navarra ( Site 0122), Madrid
- Taiwan (6):
  - Chang Gung Medical Foundation - Kaohsiung ( Site 0145), Kaohsiung City
  - China Medical University Hospital ( Site 0144), Taichung
  - National Cheng Kung University Hospital ( Site 0142), Tainan
  - National Taiwan University Hospital ( Site 0141), Taipei
  - Mackay Memorial Hospital ( Site 0143), Taipei
  - Chang Gung Memorial Hospital - Linkou Branch ( Site 0146), Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Deng JZ, Rustandi RR, Barbacci D, Swartz AR, Gulasarian A, Loughney JW. Reverse-Phase Ultra-Performance Chromatography Method for Oncolytic Coxsackievirus Viral Protein Separation and Empty to Full Capsid Quantification. Hum Gene Ther. 2022 Jul;33(13-14):765-775. doi: 10.1089/hum.2022.013. Epub 2022 Jun 1. PMID 35387488
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 76 participants were allocated and 75 participants received study intervention. The study was terminated before any participants were enrolled into Cohorts D and E.
Groups:
- Part 1, Cohort A: Triple-Negative Breast Cancer: Participants with triple-negative breast cancer (TNBC) solid tumors received 3 X 10^8 50% tissue culture infectious dose (TCID50) of gebasaxturev intratumorally for 8 cycles, and pembrolizumab intravenously for a maximum of 35 cycles. Cycle 1 was 28 days, and cycles 2-35 were 21 days.
- Part 1, Cohort B: Head and Neck Squamous Cell Carcinoma: Participants with head and neck squamous cell carcinoma (HNSCC) solid tumors received 3 X 10^8 TCID50 of gebasaxturev intratumorally for 8 cycles, and pembrolizumab intravenously for a maximum of 35 cycles. Cycle 1 was 28 days, and cycles 2-35 were 21 days.
- Part 1, Cohort C: Cutaneous Squamous Cell Carcinoma: Participants with cutaneous squamous cell carcinoma (cSCC) solid tumors received 3 X 10^8 TCID50 of gebasaxturev intratumorally for 8 cycles, and pembrolizumab intravenously for a maximum of 35 cycles. Cycle 1 was 28 days, and cycles 2-35 were 21 days.
- Part 2 Dose Level 1, Solid Tumors + Liver Metastases: Participants with solid tumors with liver metastases received 3 X 10^7 TCID50 of gebasaxturev intratumorally for 8 cycles, and pembrolizumab intravenously for a maximum of 35 cycles. Cycle 1 was 28 days, and cycles 2-35 were 21 days.
- Part 2 Dose Level 2, Solid Tumors + Liver Metastases: Participants with solid tumors with liver metastases received 1 X 10^8 TCID50 of gebasaxturev intratumorally for 8 cycles, and pembrolizumab intravenously for a maximum of 35 cycles. Cycle 1 was 28 days, and cycles 2-35 were 21 days.
- Part 2 Dose Level 3, Solid Tumors + Liver Metastases: Participants with solid tumors with liver metastases received 3 X 10^8 TCID50 of gebasaxturev intratumorally for 8 cycles, and pembrolizumab intravenously for a maximum of 35 cycles. Cycle 1 was 28 days, and cycles 2-35 were 21 days.
- Part 2, Cohort D: Hepatocellular Carcinoma (HCC): Participants with hepatocellular carcinoma (HCC) solid tumors received the gebasaxturev recommended phase 2 dose (RP2D) intratumorally for 8 cycles, and pembrolizumab intravenously for a maximum of 35 cycles. Cycle 1 was 28 days, and cycles 2-35 were 21 days. No participants were enrolled into this arm.
- Part 2, Cohort E: Gastric Carcinoma: Participants with gastric carcinoma solid tumors received the gebasaxturev recommended phase 2 dose (RP2D) intratumorally for 8 cycles, and pembrolizumab intravenously for a maximum of 35 cycles. Cycle 1 was 28 days, and cycles 2-35 were 21 days. No participants were enrolled into this arm.
Period: Overall Study
Arm/Group | Part 1, Cohort A: Triple-Negative Breast Cancer | Part 1, Cohort B: Head and Neck Squamous Cell Carcinoma | Part 1, Cohort C: Cutaneous Squamous Cell Carcinoma | Part 2 Dose Level 1, Solid Tumors + Liver Metastases | Part 2 Dose Level 2, Solid Tumors + Liver Metastases | Part 2 Dose Level 3, Solid Tumors + Liver Metastases | Part 2, Cohort D: Hepatocellular Carcinoma (HCC) | Part 2, Cohort E: Gastric Carcinoma
Started | 22 | 14 | 17 | 6 | 3 | 14 | 0 | 0
Treated | 21 | 14 | 17 | 6 | 3 | 14 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 22 | 14 | 17 | 6 | 3 | 14 | 0 | 0
Not completed — Death | 17 | 8 | 8 | 5 | 2 | 7 | 0 | 0
Not completed — Study Terminated by Sponsor | 4 | 6 | 8 | 0 | 1 | 7 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Allocated in error without study intervention | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: No participants were enrolled in Part 2 Cohort D or Part 2 Cohort E arms due to early study termination.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1, Cohort A: Triple-Negative Breast Cancer | Part 1, Cohort B: Head and Neck Squamous Cell Carcinoma | Part 1, Cohort C: Cutaneous Squamous Cell Carcinoma | Part 2 Dose Level 1, Solid Tumors + Liver Metastases | Part 2 Dose Level 2, Solid Tumors + Liver Metastases | Part 2 Dose Level 3, Solid Tumors + Liver Metastases | Total
Number analyzed (Participants) | 22 | 14 | 17 | 6 | 3 | 14 | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.5 (11.5) | 59.7 (13.1) | 80.6 (12.8) | 54.7 (12.5) | 58.3 (8.3) | 57.8 (14.1) | 62.4 (15.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 2 | 6 | 3 | 2 | 10 | 45
  Male | 0 | 12 | 11 | 3 | 1 | 4 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 0 | 0 | 0 | 0 | 0 | 4
  Not Hispanic or Latino | 18 | 14 | 13 | 6 | 3 | 11 | 65
  Unknown or Not Reported | 0 | 0 | 4 | 0 | 0 | 3 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 7 | 0 | 1 | 2 | 4 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 20 | 7 | 14 | 5 | 1 | 8 | 55
  More than one race | 2 | 0 | 0 | 0 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 3 | 0 | 0 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Objective Response Rate (ORR) Per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 as Assessed by Investigator
Description: ORR was defined as the percentage of participants in the analysis population who had a Complete Response (CR: Disappearance of all target lesions and no new lesions) or a Partial Response (PR: ≥30% decrease in the sum of diameters of target lesions) per RECIST 1.1 as assessed by investigator. For this study, RECIST 1.1 has been modified to follow a maximum of 10 target lesions and a maximum of 5 target lesions per organ, and to specify that intratumoral injection does not render a lesion non-evaluable. Per protocol, only participants in Part 1 were analyzed in this outcome measure.
Time Frame: Up to approximately 30 months
Population: The analysis population consisted of all allocated participants in Part 1 with a baseline scan that demonstrated measurable disease and who received at least 1 dose of study intervention. Cohorts D and E in Part 2 did not enroll any participants.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part 1, Cohort A: Triple-Negative Breast Cancer | Part 1, Cohort B: Head and Neck Squamous Cell Carcinoma | Part 1, Cohort C: Cutaneous Squamous Cell Carcinoma | Part 2 Dose Level 1, Solid Tumors + Liver Metastases | Part 2 Dose Level 2, Solid Tumors + Liver Metastases | Part 2 Dose Level 3, Solid Tumors + Liver Metastases
Number analyzed (Participants) | 21 | 14 | 17 | 0 | 0 | 0
Percentage of Participants | 0.0 [0.0 to 16.1] | 35.7 [12.8 to 64.9] | 64.7 [38.3 to 85.8] |  |  |

2. Primary Outcome: Number of Participants Who Experienced a Dose-Limiting Toxicity (DLT)
Description: The following toxicities during DLT evaluation period were considered a DLT, if assessed by investigator to be possibly, probably, or definitely related to treatment: Grade (Gr) 4 nonhematologic toxicity; Gr 4 hematologic toxicity lasting ≥7 days, except Gr 3 thrombocytopenia (if associated with clinically significant bleeding) or any grade febrile neutropenia; nonhematologic adverse event (AE) ≥ Gr 3 (with exceptions); Gr 3 or 4 nonhematologic lab abnormality (if medical intervention is required, leads to hospitalization, or persists for >1 week); drug-related toxicity that causes a >2 week delay in Cycle 2 initiation; drug-related toxicity that causes treatment discontinuation or missed dosage of gebasaxturev; or Gr 5 toxicity. Per protocol, only the participants in Part 2 were analyzed in this outcome measure.
Time Frame: Cycle 1 (28-day cycle)
Population: The analysis population included all allocated participants in Part 2 who received at least 1 dose of study treatment who met the criteria for DLT evaluability (e.g. finished Cycle 1 without a DLT or experienced a DLT in Cycle 1). Cohorts D and E in Part 2 did not enroll any participants.
Measure: Count of Participants; unit: Participants
Groups:
- Part 1, Cohort A: Triple-Negative Breast Cancer: Participants with triple-negative breast cancer (TNBC) solid tumors. Participants received 3 X 10^8 50% tissue culture infectious dose (TCID50) of gebasaxturev intratumorally for 8 cycles, and pembrolizumab intravenously for a maximum of 35 cycles. Cycle 1 was 28 days, and cycles 2-35 were 21 days.
Arm/Group | Part 1, Cohort A: Triple-Negative Breast Cancer | Part 1, Cohort B: Head and Neck Squamous Cell Carcinoma | Part 1, Cohort C: Cutaneous Squamous Cell Carcinoma | Part 2 Dose Level 1, Solid Tumors + Liver Metastases | Part 2 Dose Level 2, Solid Tumors + Liver Metastases | Part 2 Dose Level 3, Solid Tumors + Liver Metastases
Number analyzed (Participants) | 0 | 0 | 0 | 6 | 3 | 14
Participants |  |  |  | 1 | 0 | 1

3. Primary Outcome: Part 2: Number of Participants Who Experienced One or More Adverse Events (AEs)
Description: An AE is defined as any unfavorable and unintended sign, symptom, disease, or worsening of preexisting condition temporally associated with study treatment and irrespective of causality to study treatment. Per protocol, only participants in Part 2 were analyzed in this outcome measure.
Time Frame: Up to approximately 29 months
Population: The analysis population included all allocated participants in Part 2 who received study intervention. Cohorts D and E in Part 2 did not enroll any participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1, Cohort A: Triple-Negative Breast Cancer | Part 1, Cohort B: Head and Neck Squamous Cell Carcinoma | Part 1, Cohort C: Cutaneous Squamous Cell Carcinoma | Part 2 Dose Level 1, Solid Tumors + Liver Metastases | Part 2 Dose Level 2, Solid Tumors + Liver Metastases | Part 2 Dose Level 3, Solid Tumors + Liver Metastases
Number analyzed (Participants) | 0 | 0 | 0 | 6 | 3 | 14
Participants |  |  |  | 6 | 2 | 14

4. Primary Outcome: Part 2: Number of Participants Who Discontinued Study Intervention Due to an AE
Description: An AE was defined as any unfavorable and unintended sign, symptom, disease, or worsening of preexisting condition temporally associated with study treatment and irrespective of causality to study treatment. Per protocol, only participants in Part 2 were analyzed in this outcome measure.
Time Frame: Up to approximately 10 months
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1, Cohort A: Triple-Negative Breast Cancer | Part 1, Cohort B: Head and Neck Squamous Cell Carcinoma | Part 1, Cohort C: Cutaneous Squamous Cell Carcinoma | Part 2 Dose Level 1, Solid Tumors + Liver Metastases | Part 2 Dose Level 2, Solid Tumors + Liver Metastases | Part 2 Dose Level 3, Solid Tumors + Liver Metastases
Number analyzed (Participants) | 0 | 0 | 0 | 6 | 3 | 14
Participants |  |  |  | 0 | 0 | 1

5. Secondary Outcome: Part 1: Number of Participants Who Experienced One or More AEs
Description: An AE was defined as any unfavorable and unintended sign, symptom, disease, or worsening of preexisting condition temporally associated with study treatment and irrespective of causality to study treatment. Per protocol, only participants in Part 1 were analyzed in this outcome measure.
Time Frame: Up to approximately 30 months
Population: The analysis population included all allocated participants in Part 1 who received study intervention. Cohorts D and E in Part 2 did not enroll any participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1, Cohort A: Triple-Negative Breast Cancer | Part 1, Cohort B: Head and Neck Squamous Cell Carcinoma | Part 1, Cohort C: Cutaneous Squamous Cell Carcinoma | Part 2 Dose Level 1, Solid Tumors + Liver Metastases | Part 2 Dose Level 2, Solid Tumors + Liver Metastases | Part 2 Dose Level 3, Solid Tumors + Liver Metastases
Number analyzed (Participants) | 21 | 14 | 17 | 0 | 0 | 0
Participants | 19 | 14 | 17 |  |  |

6. Secondary Outcome: Part 1: Number of Participants Who Discontinued Study Intervention Due to an AE
Description: as for outcome 5
Time Frame: Up to approximately 23 months
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1, Cohort A: Triple-Negative Breast Cancer | Part 1, Cohort B: Head and Neck Squamous Cell Carcinoma | Part 1, Cohort C: Cutaneous Squamous Cell Carcinoma | Part 2 Dose Level 1, Solid Tumors + Liver Metastases | Part 2 Dose Level 2, Solid Tumors + Liver Metastases | Part 2 Dose Level 3, Solid Tumors + Liver Metastases
Number analyzed (Participants) | 21 | 14 | 17 | 0 | 0 | 0
Participants | 1 | 3 | 3 |  |  |

7. Secondary Outcome: Progression-Free Survival (PFS) Per RECIST 1.1 as Assessed by Investigator
Description: PFS was defined as the time from first dose of study treatment to the first documented progressive disease (PD) or death due to any cause, whichever occurs first as assessed by investigator. Per RECIST 1.1, PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD. For this study, RECIST 1.1 has been modified to follow a maximum of 10 target lesions and a maximum of 5 target lesions per organ, and to specify that intratumoral injection does not render a lesion non-evaluable. Per protocol, only participants in Part 1 were analyzed in this outcome measure.
Time Frame: Up to approximately 30 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 1, Cohort A: Triple-Negative Breast Cancer | Part 1, Cohort B: Head and Neck Squamous Cell Carcinoma | Part 1, Cohort C: Cutaneous Squamous Cell Carcinoma | Part 2 Dose Level 1, Solid Tumors + Liver Metastases | Part 2 Dose Level 2, Solid Tumors + Liver Metastases | Part 2 Dose Level 3, Solid Tumors + Liver Metastases
Number analyzed (Participants) | 21 | 14 | 17 | 0 | 0 | 0
Months | 2.1 [1.5 to 3.1] | 3.3 [1.7 to NA] — NA = Upper limit not reached at time of data cut-off due to insufficient number of participants with an event. | 15.4 [2.4 to NA] — NA = Upper limit not reached at time of data cut-off due to insufficient number of participants with an event. |  |  |

8. Secondary Outcome: Duration of Response (DOR) Per RECIST 1.1 as Assessed by Investigator
Description: For participants who demonstrated a confirmed Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: ≥30% decrease in the sum of diameters of target lesions) per RECIST 1.1 as assessed by investigator, DOR was defined as the time from first documented evidence of CR or PR until disease progression or death, whichever occurs first. For this study, RECIST 1.1 was modified to follow a maximum of 10 target lesions and a maximum of 5 target lesions per organ, and to specify that intratumoral injection did not render a lesion non-evaluable. Per protocol, only participants in Part 1 were analyzed in this outcome measure.
Time Frame: Up to approximately 30 months
Population: The analysis population consisted of all allocated participants in Part 1 who experienced a confirmed CR or PR with a baseline scan that demonstrated measurable disease and who received at least 1 dose of study intervention. No participants in Part 1, Cohort A were eligible for analysis. Cohorts D and E in Part 2 did not enroll any participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 1, Cohort A: Triple-Negative Breast Cancer | Part 1, Cohort B: Head and Neck Squamous Cell Carcinoma | Part 1, Cohort C: Cutaneous Squamous Cell Carcinoma | Part 2 Dose Level 1, Solid Tumors + Liver Metastases | Part 2 Dose Level 2, Solid Tumors + Liver Metastases | Part 2 Dose Level 3, Solid Tumors + Liver Metastases
Number analyzed (Participants) | 0 | 5 | 11 | 0 | 0 | 0
Months |  | NA [4.4 to NA] — NA = Median and upper limit not reached at time of data cut-off due to insufficient number of responding participants with relapse. | NA [4.6 to NA] — NA = Median and upper limit not reached at time of data cut-off due to insufficient number of responding participants with relapse. |  |  |

9. Secondary Outcome: PFS Per Response Evaluation Criteria in Solid Tumors 1.1 for Immune-Based Therapeutics (iRECIST) as Assessed by Investigator
Description: PFS was defined as the time from first dose of study treatment to the first documented immune-based confirmed progressive disease (iCPD) or death due to any cause, whichever occurs first as assessed by investigator. Per iRECIST, iCPD was defined as worsening of any existing cause of progression, or the appearance of any other cause of progression, relative to the initial appearance of progressive disease by RECIST 1.1. Per protocol, only participants in Part 1 were analyzed in this outcome measure.
Time Frame: Up to approximately 30 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 1, Cohort A: Triple-Negative Breast Cancer | Part 1, Cohort B: Head and Neck Squamous Cell Carcinoma | Part 1, Cohort C: Cutaneous Squamous Cell Carcinoma | Part 2 Dose Level 1, Solid Tumors + Liver Metastases | Part 2 Dose Level 2, Solid Tumors + Liver Metastases | Part 2 Dose Level 3, Solid Tumors + Liver Metastases
Number analyzed (Participants) | 21 | 14 | 17 | 0 | 0 | 0
Months | 3.3 [1.3 to 4.3] | 8.2 [2.1 to NA] — NA = Upper limit not reached at time of data cut-off due to insufficient number of participants with an event. | 20.4 [3.3 to NA] — NA = Upper limit not reached at time of data cut-off due to insufficient number of participants with an event. |  |  |

10. Secondary Outcome: DOR Per iRECIST as Assessed by Investigator
Description: For participants who demonstrated confirmed CR (disappearance of all target lesions and non-target lesions) or PR (≥30% decrease in the sum of diameters of target lesions) per RECIST 1.1 or immune-based Complete Response (iCR: Disappearance of all target lesions) or immune-based Partial Response (iPR: ≥30% decrease in the sum of diameters of target lesions) after a single PD per iRECIST, DOR was defined as the time from the first documented CR or PR, or iCR or an iPR, as assessed by investigator, until progressive disease or death, whichever occurs first. For this study, RECIST 1.1 was modified to follow a maximum of 10 target lesions and a maximum of 5 target lesions per organ, and to specify that intratumoral injection did not render a lesion non-evaluable. Per protocol, only participants in Part 1 were analyzed in this outcome measure.
Time Frame: Up to approximately 30 months
Population: The analysis population consisted of all allocated participants in Part 1 who experienced a confirmed response (CR, PR, iCR or iPR) with a baseline scan that demonstrated measurable disease and who received at least 1 dose of study intervention. No participants in Part 1, Cohort A were eligible for analysis. Cohorts D and E in Part 2 did not enroll any participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 1, Cohort A: Triple-Negative Breast Cancer | Part 1, Cohort B: Head and Neck Squamous Cell Carcinoma | Part 1, Cohort C: Cutaneous Squamous Cell Carcinoma | Part 2 Dose Level 1, Solid Tumors + Liver Metastases | Part 2 Dose Level 2, Solid Tumors + Liver Metastases | Part 2 Dose Level 3, Solid Tumors + Liver Metastases
Number analyzed (Participants) | 0 | 6 | 11 | 0 | 0 | 0
Months |  | NA [4.4 to NA] — NA = Median and upper limit not reached at time of data cut-off due to insufficient number of responding participants with relapse. | NA [4.6 to NA] — NA = Median and upper limit not reached at time of data cut-off due to insufficient number of responding participants with relapse. |  |  |

11. Secondary Outcome: ORR Per iRECIST as Assessed by Investigator
Description: ORR was defined as the percentage of participants who had confirmed responses assessed using RECIST 1.1 before PD or an immune-based Complete Response (iCR: Disappearance of all target lesions) or an immune-based Partial Response (iPR: ≥30% decrease in the sum of diameters of target lesions) after a single PD per iRECIST as assessed by investigator.
Time Frame: Up to approximately 30 months
Population: The analysis population consisted of all participants with a baseline scan that demonstrated measurable disease and who were administered at least one dose of study intervention. Cohorts D and E in Part 2 did not enroll any participants.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part 1, Cohort A: Triple-Negative Breast Cancer | Part 1, Cohort B: Head and Neck Squamous Cell Carcinoma | Part 1, Cohort C: Cutaneous Squamous Cell Carcinoma | Part 2 Dose Level 1, Solid Tumors + Liver Metastases | Part 2 Dose Level 2, Solid Tumors + Liver Metastases | Part 2 Dose Level 3, Solid Tumors + Liver Metastases
Number analyzed (Participants) | 21 | 14 | 17 | 6 | 3 | 14
Percentage of Participants | 0.0 [0.0 to 16.1] | 42.9 [17.7 to 71.1] | 64.7 [38.3 to 85.8] | 16.7 [0.4 to 64.1] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 23.2]

12. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from first dose of study intervention to death due to any cause. Per protocol, only participants in Part 1 were analyzed in this outcome measure.
Time Frame: Up to approximately 30 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 1, Cohort A: Triple-Negative Breast Cancer | Part 1, Cohort B: Head and Neck Squamous Cell Carcinoma | Part 1, Cohort C: Cutaneous Squamous Cell Carcinoma | Part 2 Dose Level 1, Solid Tumors + Liver Metastases | Part 2 Dose Level 2, Solid Tumors + Liver Metastases | Part 2 Dose Level 3, Solid Tumors + Liver Metastases
Number analyzed (Participants) | 21 | 14 | 17 | 0 | 0 | 0
Months | 7.5 [4.3 to 15.0] | 11.8 [3.0 to NA] — NA = Upper limit not reached at time of data cut-off due to insufficient number of participants with an event. | 20.4 [3.3 to NA] — NA = Upper limit not reached at time of data cut-off due to insufficient number of participants with an event. |  |  |

13. Secondary Outcome: Part 2: ORR Per RECIST 1.1 as Assessed by Investigator
Description: ORR was defined as the percentage of participants in the analysis population who had a Complete Response (CR: Disappearance of all target lesions and no new lesions) or a Partial Response (PR: ≥30% decrease in the sum of diameters of target lesions) per RECIST 1.1 as assessed by investigator. For this study, RECIST 1.1 was modified to follow a maximum of 10 target lesions and a maximum of 5 target lesions per organ, and to specify that intratumoral injection does not render a lesion non-evaluable. Per protocol, only participants in Part 2 were analyzed for this outcome measure.
Time Frame: Up to approximately 29 months
Population: The analysis population consisted of all allocated participants in Part 2 with a baseline scan that demonstrated measurable disease and who received at least 1 dose of study intervention. Cohorts D and E in Part 2 did not enroll any participants
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part 1, Cohort A: Triple-Negative Breast Cancer | Part 1, Cohort B: Head and Neck Squamous Cell Carcinoma | Part 1, Cohort C: Cutaneous Squamous Cell Carcinoma | Part 2 Dose Level 1, Solid Tumors + Liver Metastases | Part 2 Dose Level 2, Solid Tumors + Liver Metastases | Part 2 Dose Level 3, Solid Tumors + Liver Metastases
Number analyzed (Participants) | 0 | 0 | 0 | 6 | 3 | 14
Percentage of Participants |  |  |  | 16.7 [0.4 to 64.1] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 23.2]

ADVERSE EVENTS:
Time Frame: Up to approximately 30 months
Description: Serious and Other adverse events (AEs) includes all participants who received ≥1 dose of study drug. All-Cause Mortality includes all allocated participants. Per protocol, disease progression of cancer under study was not considered an AE unless considered related to study treatment. Thus, MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" & "Disease progression" not related to study treatment are excluded as AEs. No participants were allocated to Cohort D or E.
Arm/Group | Part 1, Cohort A: Triple-Negative Breast Cancer | Part 1, Cohort B: Head and Neck Squamous Cell Carcinoma | Part 1, Cohort C: Cutaneous Squamous Cell Carcinoma | Part 2 Dose Level 1, Solid Tumors + Liver Metastases | Part 2 Dose Level 2, Solid Tumors + Liver Metastases | Part 2 Dose Level 3, Solid Tumors + Liver Metastases
All-Cause Mortality (participants affected / at risk) | 18/22 | 8/14 | 8/17 | 5/6 | 2/3 | 7/14
Serious Adverse Events (participants affected / at risk) | 4/21 | 8/14 | 6/17 | 4/6 | 1/3 | 3/14
Other Adverse Events (participants affected / at risk) | 18/21 | 14/14 | 17/17 | 6/6 | 2/3 | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1, Cohort A: Triple-Negative Breast Cancer (N=21) | Part 1, Cohort B: Head and Neck Squamous Cell Carcinoma (N=14) | Part 1, Cohort C: Cutaneous Squamous Cell Carcinoma (N=17) | Part 2 Dose Level 1, Solid Tumors + Liver Metastases (N=6) | Part 2 Dose Level 2, Solid Tumors + Liver Metastases (N=3) | Part 2 Dose Level 3, Solid Tumors + Liver Metastases (N=14)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Liver abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic seroma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Troponin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Polyneuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lichenoid keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1, Cohort A: Triple-Negative Breast Cancer (N=21) | Part 1, Cohort B: Head and Neck Squamous Cell Carcinoma (N=14) | Part 1, Cohort C: Cutaneous Squamous Cell Carcinoma (N=17) | Part 2 Dose Level 1, Solid Tumors + Liver Metastases (N=6) | Part 2 Dose Level 2, Solid Tumors + Liver Metastases (N=3) | Part 2 Dose Level 3, Solid Tumors + Liver Metastases (N=14)
Anaemia (Blood and lymphatic system disorders) | 5 (5) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (3)
Hyperleukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deafness (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 5 (5) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 4 (4) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thyroiditis (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Exophthalmos (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Anorectal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (2) | 4 (12) | 0 (0) | 0 (0) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (8) | 2 (2) | 0 (0) | 1 (2) | 1 (1) | 5 (9)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Salivary gland pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tongue geographic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (9)
Asthenia (General disorders) | 2 (2) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 3 (5)
Chills (General disorders) | 4 (6) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 1 (1)
Discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Face oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (8) | 3 (3) | 4 (4) | 3 (3) | 0 (0) | 4 (5)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5)
Injection site bruising (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site inflammation (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 2 (5) | 1 (2) | 2 (2) | 2 (3) | 0 (0) | 2 (5)
Injection site pruritus (General disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 6 (10) | 1 (2) | 2 (2) | 2 (2) | 1 (1) | 5 (8)
Swelling face (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 5 (5) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stoma complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 4 (4) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 4 (4) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 3 (3)
Bilirubin conjugated increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Blood creatine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Blood urea increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CD4 lymphocytes increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Protein total decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thyroxine free increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thyroxine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Troponin T increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 2 (2)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (3)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 4 (4) | 0 (0) | 0 (0) | 4 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (4)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemangioma of spleen (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (6) | 2 (2) | 4 (5) | 1 (2) | 0 (0) | 3 (4)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Post herpetic neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hallucination, visual (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nocturia (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic discomfort (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Perineal pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (4) | 1 (1) | 1 (2) | 1 (1) | 3 (3)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin erosion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vitiligo (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor will generally support publication of multicenter studies only in their entirety and not as individual site data. In this case, a coordinating investigator will be designated by mutual agreement. If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-25): https://cdn.clinicaltrials.gov/large-docs/21/NCT04521621/Prot_SAP_000.pdf